CLINICAL TRIAL: NCT00057941
Title: A Randomized Phase II Trial of Combination Anastrozole (NSC #719344) Plus ZD1839 (Iressa, NSC #715055, IND #61187) and of Combination Fulvestrant (NSC #719276) Plus ZD1839 in the Treatment of Postmenopausal Women With Hormone Receptor-Positive Metastatic Breast Cancer
Brief Title: Anastrozole and ZD1839 Compared With Fulvestrant and ZD1839 in Postmenopausal Women w/ Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03148; NCI-2012-03148 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000285631; U10CA021115 (NIH); E4101 (Other: Eastern Cooperative Oncology Group); E4101 (Other: CTEP)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2013-01

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Progesterone Receptor-positive Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Gefitinib; Fulvestrant

ARMS (2):
- Arm I (anastrozole, gefitinib) (Experimental): Patients receive oral anastrozole and oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: anastrozole; Drug: gefitinib; Other: laboratory biomarker analysis
- Arm II (fulvestrant, gefitinib) (Experimental): Patients receive fulvestrant intramuscularly on day 1 and oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gefitinib; Drug: fulvestrant; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: anastrozole — Given orally
  Other Names: ANAS; Arimidex; ICI-D1033
  Arms: Arm I (anastrozole, gefitinib)
Drug: gefitinib — Given orally
  Other Names: Iressa; ZD 1839
Drug: fulvestrant — Given intramuscularly
  Other Names: Faslodex; ICI 182,780
  Arms: Arm II (fulvestrant, gefitinib)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well giving gefitinib together with anastrozole works compared to giving gefitinib together with fulvestrant in treating postmenopausal women with recurrent or metastatic breast cancer. Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using anastrozole and fulvestrant may fight breast cancer by blocking the use of estrogen. Gefitinib (ZD1839) may stop the growth of cancer cells by blocking the enzymes necessary for their growth. It is not yet known whether gefitinib is more effective when combined with anastrozole or fulvestrant in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the antitumor activity of anastrozole given in combination with the EGFR tyrosine kinase inhibitor ZD1839, and of fulvestrant given in combination with the EGFR tyrosine kinase inhibitor ZD1839.

II. Evaluate the safety of anastrozole given in combination with ZD1839 and fulvestrant given in combination with ZD1839.

III. Evaluate the interaction of biological characteristics that predict for response of breast cancer to treatment with anastrozole and ZD1839 and with fulvestrant and ZD1839.

OUTLINE: This is a randomized, open-label study. Patients are stratified according to prior hormonal therapy (yes vs. no) and dominant site of disease (soft tissue/lymph nodes vs. bone vs. visceral). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral anastrozole and oral gefitinib once daily on days 1-28.

Arm II: Patients receive fulvestrant intramuscularly on day 1 and oral gefitinib once daily on days 1-28.

Courses in both arms repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have estrogen and/or progesterone receptor positive histologically confirmed adenocarcinoma of the breast with measurable recurrent or metastatic carcinoma of the breast
* Baseline measurements and evaluations of involved sites should be performed as close as possible to study entry, but must be within 4 weeks prior to randomization
* Patients with available tissue blocks from either the primary or metastatic site must submit the tissue for EGFR analysis
* All patients must be postmenopausal females defined by:

  * Prior bilateral oophorectomy or bilateral ovarian irradiation
  * No menstrual period for 12 months or longer. If age 55 years or less and on tamoxifen within the prior 6 months, must have an estradiol level in the postmenopausal range
* Patients must not have had more than 2 prior chemotherapy regimens for metastatic disease and no chemotherapy within 3 weeks prior to randomization; no concurrent chemotherapy is allowed while on protocol therapy
* Patients must not have prior hormonal therapy for metastatic disease; no prior therapy in the adjuvant setting with an estrogen receptor down-regulator (e.g. fulvestrant) or an aromatase inhibitor (e.g. anastrozole, letrozole, exemestane, aminoglutethamide); non-protocol concurrent hormonal therapy is not allowed
* Patients must not have had prior therapy with agents that target EGFR
* Previous, but not concomitant, therapy with trastuzumab (Herceptin) is allowed; patients must not receive trastuzumab (Herceptin) within 3 weeks prior to randomization
* Patients must have ECOG performance status of 0, 1, or 2
* Neutrophils >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Bilirubin =< 1.25 x upper limit of normal
* SGPT (ALT) and SGOT (AST) =< 2.5 x upper limit of normal if no demonstrable liver metastases or =< 5 times upper limit of normal in the presence of liver metastases
* Calculated creatinine clearance >= 30ml/min
* INR, PT and PTT within normal range
* Patients must not be receiving therapy with anticoagulants or have other contraindication to i.m. injections
* Patients must not have a history of central nervous system metastasis
* Patients may receive concurrent radiation therapy to painful sites of boney disease or areas of impending fracture as long as the radiation therapy is initiated prior to study entry and sites of measurable disease outside the radiation therapy port are available to follow; patient who have received prior radiation therapy must have recovered from toxicity of the prior radiation therapy
* Patients must not take the following medications that may alter ZD1839 pharmacokinetics while enrolled in this trial: phenytoin, carbamazapine, phenobarbitol, rifampicin, and St. John's Wort, oxcarbazepine, rifapentine, modafinil, and griseofulvin
* Patients age =< 55 years must not be receiving LHRH agonists or antagonists within 3 months prior to randomization
* Patients who have an ocular inflammation or infection should be fully treated before entry into the trial; patients with a neuropathic keratopathy or diabetes or those with anterior basement membrane disease must be advised of the need for frequent opthalmalogic exams
* Patients who continue to wear contact lenses must be advised that they have an increased risk of ocular events; the decision to wear contact lenses should be discussed with the patient's treating oncologist and ophthalmologist
* Patients must not suffer from medical or psychiatric conditions that would interfere with protocol compliance, the ability to provide informed consent, or assessment of response or anticipated toxicities
* Patients must be disease-free of prior invasive malignancies for > 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2003-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Carlson, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Carlson RW, O'Neill A, Vidaurre T, Gomez HL, Badve SS, Sledge GW. A randomized trial of combination anastrozole plus gefitinib and of combination fulvestrant plus gefitinib in the treatment of postmenopausal women with hormone receptor positive metastatic breast cancer. Breast Cancer Res Treat. 2012 Jun;133(3):1049-56. doi: 10.1007/s10549-012-1997-5. Epub 2012 Mar 15. PMID 22418699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened on September 16, 2003 and closed on May 29, 2007, with final accrual of 148 patients, 74 on each arm. Patients were accrued through ECOG group.
Groups:
- Arm I (Anastrozole and ZD1839): Patients receive oral anastrozole and oral gefitinib once daily on days 1-28.
- Arm II (Fulvestrant and ZD1839): Patients receive fulvestrant intramuscularly on day 1 and oral gefitinib once daily on days 1-28.
Period: Overall Study
Arm/Group | Arm I (Anastrozole and ZD1839) | Arm II (Fulvestrant and ZD1839)
Started | 74 | 74
Treated | 74 | 74
Eligible | 72 | 69
Completed | 0 | 0
Not Completed | 74 | 74
Not completed — Death | 1 | 2
Not completed — Adverse Event | 7 | 9
Not completed — Lack of Efficacy | 54 | 53
Not completed — Withdrawal by Subject | 6 | 1
Not completed — still on treatment | 3 | 1
Not completed — insurance, symptomatic deterioration | 1 | 3
Not completed — Ineligible | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Anastrozole and ZD1839) | Arm II (Fulvestrant and ZD1839) | Total
Number analyzed (Participants) | 72 | 69 | 141
Age, Continuous [Median (Full Range); unit: years] | 58 [34 to 90] | 63 [35 to 91] | 59 [34 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 69 | 141
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78
  Peru | 33 | 29 | 62
  South Africa | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate
Description: Clinical benefit = complete response (CR), partial response (PR), or stable disease (SD) lasting for at least 6 months, assessed per Response Evaluation Criteria of Solid Tumor (RECIST).CR=disappearance of all target and non-target lesions. PR= disappearance of or at least 30% decrease in the sum of the longest diameters of target lesions, with non-progressive disease in non-target lesions. SD= sum of the longest diameters of target lesions decrease <30% or increase <20%, with non-progressive disease in non-target lesions. 141 eligible, treated patients were included.
Time Frame: assessed every 3 cycles while on treatment, assessed every 3 months when follow up <2 years, every 6 months between 2-3 years,no specific requirements after 3 years
Population: 141 eligible and treated patients, 72 on Arm I (Anastrozole and ZD1839) and 69 on Arm II (Fulvestrant and ZD1839)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anastrozole and ZD1839 | Fulvestrant and ZD1839
Number analyzed (Participants) | 72 | 69
percentage of participants | 44 [33 to 57] | 41 [29 to 53]

ADVERSE EVENTS:
Time Frame: Assessed each cycle (4 weeks) while on treatment and for 30 days after the end of treatment
Arm/Group | Arm I (Anastrozole and ZD1839) | Arm II (Fulvestrant and ZD1839)
Serious Adverse Events (participants affected / at risk) | 27/74 | 28/74
Other Adverse Events (participants affected / at risk) | 72/74 | 70/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Anastrozole and ZD1839) (N=74) | Arm II (Fulvestrant and ZD1839) (N=74)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Investigations) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Thrombosis/Embolism (Vascular disorders) | 1 | 1
Fatigue (General disorders) | 2 | 2
Weight loss (Investigations) | 0 | 1
Elevated Partial thromboplastin time (PTT) (Investigations) | 1 | 0
Elevated Prothrombin Time (PT) (Investigations) | 1 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4 | 10
Bilirubin increased (Metabolism and nutrition disorders) | 1 | 2
AST increased (Hepatobiliary disorders) | 5 | 6
ALT increased (Hepatobiliary disorders) | 3 | 3
Infection w/o neutropenia (Infections and infestations) | 1 | 3
Lymphatics-other (Infections and infestations) | 1 | 0
Joint,muscle, bone-other (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tearing (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Headache (Nervous system disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Creatinine increased (Investigations) | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Ureteral obstruction (Renal and urinary disorders) | 1 | 0
Vaginitis (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Anastrozole and ZD1839) (N=74) | Arm II (Fulvestrant and ZD1839) (N=74)
Anemia (Blood and lymphatic system disorders) | 16 | 12
Leukopenia (Investigations) | 7 | 8
Neutropenia (Investigations) | 4 | 7
Edema (General disorders) | 6 | 3
Fatigue (General disorders) | 31 | 25
Weight loss (Investigations) | 7 | 6
Elevated Partial Thromboplastin Time (PTT) (Investigations) | 9 | 10
Elevated Prothrombin Time (PT) (Investigations) | 6 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 45 | 46
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 4 | 6
Nail change (Skin and subcutaneous tissue disorders) | 6 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 18
Rash/desquamation (Skin and subcutaneous tissue disorders) | 41 | 35
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 8
Hot flashes (Vascular disorders) | 11 | 5
Anorexia (Metabolism and nutrition disorders) | 19 | 19
Constipation (Gastrointestinal disorders) | 4 | 6
Dehydration (Metabolism and nutrition disorders) | 28 | 31
Dyspepsia (Gastrointestinal disorders) | 7 | 7
Nausea (Gastrointestinal disorders) | 20 | 15
Stomatitis (Gastrointestinal disorders) | 15 | 10
Vomiting (Gastrointestinal disorders) | 12 | 9
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 37 | 38
Alkaline phosphatase increased (Investigations) | 5 | 5
Bilirubin increased (Metabolism and nutrition disorders) | 7 | 14
AST increased (Hepatobiliary disorders) | 25 | 29
ALT increased (Hepatobiliary disorders) | 26 | 26
Infection w/o neutropenia (Infections and infestations) | 8 | 7
Neuropathy-motor (Nervous system disorders) | 6 | 4
Neuropathy-sensory (Nervous system disorders) | 4 | 1
Conjunctivitis (Eye disorders) | 4 | 5
Dry eye (Eye disorders) | 5 | 6
Abdominal pain (Gastrointestinal disorders) | 9 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 11 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 9
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Pain-other (General disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Creatinine increased (Investigations) | 5 | 6
Dysuria (Renal and urinary disorders) | 5 | 2
Urinary frequency/urgency (Renal and urinary disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less